CLINICAL TRIAL: NCT00696696
Title: A Phase II Study of Gemcitabine and Erlotinib Plus Sorafenib (GES) in Metastatic Pancreatic Cancer
Brief Title: Study of Gemcitabine and Erlotinib Plus Sorafenib (GES) in Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Bayer (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYU 06-882
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Results first posted 2011-12-21 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-05

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic adenocarcinoma; metastatic; EGRF inhibitor; targeted therapy; combined cancer therapy; kinase inhibitor; VEGF-R inhibitor
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — Gemcitabine; Erlotinib Hydrochloride; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination GES (Experimental): Combination of Gemcitabine, Erlotinib, and Sorafenib
  Interventions: Drug: Gemcitabine; Drug: Erlotinib; Drug: Sorafenib

INTERVENTIONS:
Drug: Gemcitabine — 1000 mg/m^2, intravenous, Days 1, 8, 15 for every 28-day cycle. In the absence of disease progression or toxicity, a patient may continue to receive gemcitabine, erlotinib, and sorafenib until disease progression.
  Other Names: Gemzar
Drug: Erlotinib — 150 mg, taken orally, once a day, Days 1-28 for every 28-day cycle. In the absence of disease progression or toxicity, a patient may continue to receive gemcitabine, erlotinib, and sorafenib until disease progression.
  Other Names: Tarceva; OSI-774; CP-358
Drug: Sorafenib — 400 mg, taken orally, twice a day, Days 1-28 for every 28-day cycle. In the absence of disease progression or toxicity, a patient may continue to receive gemcitabine, erlotinib, and sorafenib until disease progression.
  Other Names: Nexavar; BAY 43-9006

SUMMARY:
This study tests the combination of two targeted therapies,along with chemotherapy treatment in the treatment of pancreatic cancer.

DETAILED DESCRIPTION:
Until very recently, additional therapies in pancreatic cancer have targeted either the vascular endothelial growth factor (VEGF) or epidermal growth factor (EGF) pathways, a strategy which has shown variable clinical efficacy. This inconsistency is not surprising, given the knowledge that tumors have a certain level of signal redundancy which may limit the effectiveness of any one single-targeted therapy. The dual blockade of the EGF and VEGF pathways takes aim at two of the most active cascades in tumorigenesis. Preliminarily, a phase II study done in pancreatic cancer with gemcitabine, bevacizumab and erlotinib or cetuximab has shown promising results and will most likely proceed to phase III study for definitive efficacy assessment (Kindler et al, 2006).

In this study, targeted blockade is carried one step further with the inhibition of the signaling cascade downstream of receptor tyrosine kinases at the level of raf. Given the fact that the majority of pancreatic tumors display constitutive activation of the Ras/Raf/MEK/ERK pathway, it is hoped that the addition of sorafenib to gemcitabine and erlotinib will obtain a more complete blockade of the signal transduction cascade responsible for pancreatic tumor growth and progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed pancreatic adenocarcinoma not amenable to curative treatment with surgery. Patients with locally advanced disease must have disease that extends outside the boundaries of a standard radiation port.
* Measurable disease, as defined by Response Evaluation Criteria In Solid Tumors (RECIST). This requires at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan. Pleural effusions and ascites are not considered measurable lesions.
* No prior cytotoxic chemotherapy for metastatic disease. Prior adjuvant chemotherapy is allowed, however at least 6 months must have elapsed from administration of the last dose of chemotherapy or radiotherapy.
* No prior therapy with a VEGF, EGFR, or multi-targeted kinase inhibitor.
* Age >18 years.
* Life expectancy of greater than 3 months.
* Eastern Cooperative Oncology Group performance status 0-1.
* Normal organ and marrow function as defined below:

  * White blood cells (WBC) >3,000/µl
  * Absolute neutrophil count >1,500/µl
  * Platelets >100,000/µl
  * Total bilirubin ≤ 2.5 x institutional upper limit of normal (ULN)
  * Transaminases(SGOT/ SGPT)

    * without liver mets ≤ 2.5 x institutional ULN
    * with liver mets ≤ 5 x institutional ULN
  * International Normalized Ratio (INR)

    * patients not on warfarin ≤ 1.5
    * patients on warfarin ≤ 3
  * Renal Function: Serum creatinine ≤ 1.5 xULN
  * Proteinuria: Urine protein <1+, or 24hr urine protein <500 mg
* At least 30 days since receiving any investigational drug.
* Patients who received prior radiation therapy must have a site of measurable disease that is not located within the prior radiation port.
* Patients who are on warfarin anticoagulation are allowed to participate as long as they fit the following 3 criteria:

  * They are therapeutic on a stable warfarin dose
  * Their INR target range is no greater than 3
  * They are monitored with regular INR testing
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment.
* Women of childbearing potential and men must agree to use adequate contraception (barrier method birth control) prior to study entry and for the duration of study participation. Men should use adequate birth control for at least three months after the last administration of study drugs.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* No prior treatment with bevacizumab, cetuximab, or erlotinib. Prior gemcitabine in the adjuvant setting completed more than six months previously will be allowed.
* No other investigational agents.
* No central nervous system (CNS) disease, including primary brain tumors, brain metastasis, or history of a cerebro-vascular accident (CVA) or transient ischemic attack (TIA) within 6 months of starting therapy.
* No allergic reactions to compounds similar to erlotinib or sorafenib.
* Because an increased risk of bleeding may occur following sorafenib administration, no patients will be allowed with a history of bleeding diathesis or coagulopathy. No grade > 2 pulmonary hemorrhage or > grade 3 other hemorrhage within 28 days of beginning therapy.
* No recent invasive procedures defined as follows: Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to Day 1 of therapy
* No Patients with clinically significant cardiovascular disease, defined as:

  * Uncontrolled hypertension
  * Myocardial infarction < 6 months prior to registration and new onset angina within 3 months (controlled stable angina acceptable)
  * New York heart association grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, unstable angina pectoris
  * Grade II or greater peripheral vascular disease
* No serious or non-healing wound, ulcer, or bone fracture.
* No active infection requiring parental antibiotics.
* No currently active second malignancy other than non-melanoma skin cancer or carcinoma in-situ of the cervix.
* If a patient is on full-dose anticoagulants (warfarin or low molecular weight heparins are allowed), the following criteria should be met for enrollment: they must have a therapeutic INR, no greater than 3, on a stable dose of warfarin.
* No use of thrombolytic agents within 1 month of study initiation.
* No gastrointestinal tract disease resulting in an inability to take oral medication or prior surgical procedures affecting absorption. This may include patients with or without requirements for IV alimentation.
* No women who are pregnant (positive pregnancy test) or nursing. Fertile men and women must agree to use adequate contraceptive measures during study therapy and for at least 3 months after the completion of antibody therapy.
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, no HIV-positive patients, including those receiving combination anti-retroviral therapy, are allowed on the study.
* Any condition that impairs patient's ability to swallow whole pills
* Any malabsorption problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-09; Primary Completion 2010-11 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Cohen, MD, Principal Investigator — NYU School of Medicine
Locations (3):
- United States (3):
  - Desert Regional Medical Center, Palm Springs, California
  - Bellevue Hospital, New York, New York
  - New York University Cancer Center, New York, New York

REFERENCES:
- [Background] Kindler HL, K. A. Bylow, H. S. Hochster, G. Friberg, K. Micetich, G. Locker, M. Kozloff, M. Moore, W. Sun, E. E. Vokes, and University Of Chicago Phase II Consortium. A randomized phase II study of bevacizumab (B) and gemcitabine (G) plus cetuximab (C) or erlotinib (E) in patients with advanced pancreatic cancer: A preliminary analysis. J. Clin. Oncol (Meeting Abstracts) June 2006, vol. 24 no. 18_suppl 4040
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled 45 patients from September 2007 to May 2010 at New York University Medical center and affiliated hospital, New York, NY and Desert Regional Medical center, Palm Springs, CA.
Pre-assignment Details: One patient was enrolled but then withdrew consent before treatment.
Period: Overall Study
Arm/Group | Combination GES
Started | 44
Completed | 26 (number of patients off treatment due to progression of disease only)
Not Completed | 18
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 8
Not completed — Physician Decision | 2
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | Combination GES
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 22
Age, Continuous [Median (Full Range); unit: years] | 64 (9) [45 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: 4-month Progression Free Survival (PFS) Rate
Description: The PFS rate at 4 months is defined as the percentage of patients whose disease is progression free at 4 months from the start of treatment. Disease progression is evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) (Therasse et al, 2000). Radiological measurements to determine progression is performed every 2 cycles.
Time Frame: 4 months
Population: Based on the number of patients treated.
Measure: Number; unit: percentage of patients
Arm/Group | Combination GES
Number analyzed (Participants) | 44
percentage of patients | 49

2. Secondary Outcome: Objective Response Rate
Description: The response rate is the percentage of the patients who have a complete response or partial response based on RECIST from the start of the treatment. The response is evaluated every 2 cycles by radiologic methods (e.g., computer tomography (CT)).
Time Frame: up to 1 year
Population: Based on the number of patients evaluable for response. The evaluable patients were those patients who received any treatment and had first response assessment followed by at least one confirmatory scan.
Measure: Number; unit: percentage of patients
Arm/Group | Combination GES
Number analyzed (Participants) | 30
percentage of patients | 7

3. Secondary Outcome: Median Overall Survival (mOS)
Description: Median overall survival is defined as the time when 50% of the patients are alive from the start of the treatment.
Time Frame: up to 2 years
Population: Based on the number of patients treated.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Combination GES
Number analyzed (Participants) | 44
days | 195 [144 to 290]

ADVERSE EVENTS:
Time Frame: up to 1 year (treatment period plus 30 days after the treatment)
Description: All the events were included regardless they were related or not related to the treatment drugs.
Arm/Group | Combination GES
Serious Adverse Events (participants affected / at risk) | 14/44
Other Adverse Events (participants affected / at risk) | 36/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination GES (N=44)
AST, SGOT (Investigations) | 1 (1)
anorexia (Gastrointestinal disorders) | 1 (1)
bilirubin (Investigations) | 1 (1)
cardiac general (Cardiac disorders) | 1 (1)
confusion (Nervous system disorders) | 1 (1)
constitutional symptoms (General disorders) | 2 (4)
diarrhea (Gastrointestinal disorders) | 2 (2)
febrile neutropenia (Infections and infestations) | 1 (1)
fever (General disorders) | 1 (1)
hemorrhage (GI) (Gastrointestinal disorders) | 1 (1)
hypotension (Cardiac disorders) | 1 (1)
infection with normal Anc or grade 1 or 2 neutropenia (Infections and infestations) | 1 (1)
infection with unknown Anc (Infections and infestations) | 1 (2)
nausea (Gastrointestinal disorders) | 1 (1)
obstruction (Gastrointestinal disorders) | 1 (2)
perforation (Gastrointestinal disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination GES (N=44)
albumin, serum-low (hypoalbuminemia) (Investigations) | 8 (18)
alkaline phosphatase (Investigations) | 10 (14)
anorexia (Gastrointestinal disorders) | 13 (21)
bicarbonate, serum-low (Metabolism and nutrition disorders) | 5 (7)
bilirubin (hyperbilirubinemia) (Investigations) | 4 (8)
blood/bone marrow-other (Blood and lymphatic system disorders) | 10 (25)
bruising (Skin and subcutaneous tissue disorders) | 2 (3)
constipation (Gastrointestinal disorders) | 4 (5)
constitutional symptons-other (General disorders) | 2 (2)
dermatology/skin-other (Skin and subcutaneous tissue disorders) | 10 (18)
diarrhea (Gastrointestinal disorders) | 25 (54)
distension/bloating, abdominal (Gastrointestinal disorders) | 12 (22)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
edema: limb (Blood and lymphatic system disorders) | 6 (11)
fatigue (General disorders) | 21 (36)
febrile neutropenia (fever of unknown origin without clinically or microbiologically documentation (Infections and infestations) | 3 (7)
fever (in the absence of neutropenia) (General disorders) | 7 (13)
flatulence (Gastrointestinal disorders) | 5 (12)
hair loss/alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
hemoglobin (Blood and lymphatic system disorders) | 14 (25)
hemorrhage (GI) (Gastrointestinal disorders) | 4 (5)
hemorrhage (pulmonary/upper respiratory) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
hemorrhage/bleeding-other (General disorders) | 5 (10)
hemorrhoid (Gastrointestinal disorders) | 2 (3)
hiccoughs (Respiratory, thoracic and mediastinal disorders) | 2 (2)
hypocalcemia (Metabolism and nutrition disorders) | 4 (9)
hyperglycemia (Metabolism and nutrition disorders) | 6 (9)
hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
hypernatremia (Metabolism and nutrition disorders) | 2 (2)
hypertension (Cardiac disorders) | 2 (2)
hypokalemia (Metabolism and nutrition disorders) | 4 (4)
hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
hyponatremia (Metabolism and nutrition disorders) | 4 (6)
infection with normal Anc or grade 1 or 2 neutrophils (Infections and infestations) | 2 (2)
infection-other (Infections and infestations) | 2 (2)
insomnia (General disorders) | 3 (3)
leukocytes (Blood and lymphatic system disorders) | 10 (35)
lymphopenia (Blood and lymphatic system disorders) | 8 (27)
metabolic/laboratory-other (General disorders) | 3 (3)
mood alteration (Nervous system disorders) | 3 (4)
mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 4 (4)
mucositis/stomatits (clinical exam) (Gastrointestinal disorders) | 2 (2)
nail changes (Skin and subcutaneous tissue disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 13 (36)
neuropathy: sensory (Nervous system disorders) | 2 (2)
neutrophils/granulocytes (Blood and lymphatic system disorders) | 6 (18)
pain (General disorders) | 21 (42)
pain-other (General disorders) | 4 (5)
petechiae/purpura (Skin and subcutaneous tissue disorders) | 2 (2)
pulmonary/upper respiratory-other (Respiratory, thoracic and mediastinal disorders) | 2 (3)
rash/desquamation (Skin and subcutaneous tissue disorders) | 10 (13)
rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 17 (32)
rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 12 (22)
rigors/chills (General disorders) | 8 (10)
serum glutamic oxaloacetic transaminase (ALT/SGOT) (Investigations) | 8 (9)
serum glutamic pyruvic transaminase (AST/SGPT) (Investigations) | 7 (9)
skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
sweating (diaphoresis) (General disorders) | 2 (5)
syndromes-other (General disorders) | 4 (4)
taste alteration (dysgeusia) (Gastrointestinal disorders) | 3 (3)
thrombosis/thrombus/embolism (Vascular disorders) | 2 (2)
vision-blurred vision (Eye disorders) | 2 (2)
voice changes (Respiratory, thoracic and mediastinal disorders) | 3 (4)
vomiting (Gastrointestinal disorders) | 11 (21)
weight loss (General disorders) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No